CLINICAL TRIAL: NCT04032184
Title: Effectiveness of Different Preventive Regimens in Cariogram Parameters and DMF Scores of High Caries Risk Patients: A Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Howaida Fakhry Fouad, Resident of conservative departement , Faculty of Oral and Dental Medicine, Cairo university 2012, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1234567
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Prevention of Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluoride toothpaste (Active Comparator)
  Interventions: Other: Fluoride toothpaste
- fluoride toothpaste and chlorhexidine mouthwash (Experimental)
  Interventions: Other: fluoride toothpaste and chlorhexidine mouthwash
- fluoride toothpaste, chlorhexidine mouthwash, MI varnish (Experimental)
  Interventions: Other: fluoride toothpaste, chlorhexidine mouthwash, MI varnish

INTERVENTIONS:
Other: Fluoride toothpaste — regimen using fluoride toothpaste
  Arms: Fluoride toothpaste
Other: fluoride toothpaste and chlorhexidine mouthwash — regimen using fluoride toothpaste and chlorhexidine mouthwash
  Arms: fluoride toothpaste and chlorhexidine mouthwash
Other: fluoride toothpaste, chlorhexidine mouthwash, MI varnish — regimen using fluoride toothpaste, chlorhexidine mouthwash, MI varnish
  Arms: fluoride toothpaste, chlorhexidine mouthwash, MI varnish

SUMMARY:
66 Participants will be divided into three groups according to the tested regimen (A), where (A1) represents participants exposed to fluoride toothpaste, (A2) represents participants exposed to regimen including fluoride toothpaste and chlorhexidine mouthwash and (A3) represents participants exposed to regimen including fluoride toothpaste, chlorhexidine mouthwash and MI fluoride varnish. The study will be carried over a period of one year, assessment of cariogram will be done in two visits: first visit (baseline: T0) and second visit (after 3 months: T2). In addition assessment of DMF scores will be done in four visits: first visit (baseline: T0), second visit (after 3 months: T1), third visit (after 6 months: T2) and final visit (after 12 months: T3) to obtain the required data

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-50 years
* High caries risk patients defined according to cariogram caries risk assessment model
* On non-cariogenic diet
* High plaque index
* Systematically healthy
* No orthodontic or prosthodontic appliance

Exclusion Criteria:

* Age range less than 20 or more than 50 years
* Low or moderate caries risk patients according to cariogram
* Patients with a compromised medical history
* Cariogenic diet patient
* Participants with a history of allergy to any of the drugs or chemicals used in the study
* Patients on any antibiotics during the past month

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Caries Risk Assessment | an average 3 months
  will be evaluated by cariogram

SECONDARY OUTCOMES:
DMF scores | an average of 12 months
  will be evaluated by ICDAS

CONTACTS AND LOCATIONS:
Locations (1):
- Howaida Fakhry Fouad, Giza, Other, Egypt

IPD SHARING:
Plan to Share IPD: Undecided